CLINICAL TRIAL: NCT06616779
Title: An Open, Single-centre, Non-interventional Study of the CE-marked Medical Device GlucoTab, According to Intended Use Without Additional Invasive and Stressful Measures
Brief Title: DigiDiab Evaluation Domiciliary Nursing Care
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: DigiDiab Styria
Record Dates: First submitted 2024-09-19; First posted 2024-09-27 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes; Type 2 Diabetes Mellitus (T2DM); Type 2 Diabetes, Insulin Requiring
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GlucoTab Group
  Interventions: Device: GlucoTab
- Retrospective Control Group
  Interventions: Other: Diabetes Treatment

INTERVENTIONS:
Device: GlucoTab — Insulin therapy will be started and adjusted according to the GlucoTab system with incorporated software algorithm. The goal of the basal insulin algorithm is to maintain blood glucose (BG) within acceptable targets according to the predefined health status. For a limited time period after therapy start, three BG measurements per day are suggested by the algorithm to determine blood glucose. Insulin dosage titration will be performed according to the algorithm in GlucoTab under supervision of the nurses of domiciliary nursing care. Correctional bolus insulin will be administered at defined time-points according to BG targets in the predefined health status. Nurses and nursing assistants will be trained in the use of the GlucoTab system.
  Groups: GlucoTab Group
Other: Diabetes Treatment — Diabetes Standard Care
  Groups: Retrospective Control Group

SUMMARY:
GlucoTab is a stand-alone software system to support healthcare professionals in the care of patients with diabetes mellitus or newly diagnosed hyperglycaemia who are treated with insulin and/or other glucose-lowering drugs or of patients only requiring glucose monitoring.

It provides a therapy algorithm for subcutaneous basal insulin therapy of patients with type 2 diabetes, which will be used in this study.

DETAILED DESCRIPTION:
GlucoTab: The CE-marked medical device GlucoTab is a system designed to support healthcare personnel in managing insulin therapy for patients with diabetes.

In this study, only the GlucoTab algorithm supported basal therapy will be used, which is intended for patients with Type 2 diabetes in domiciliary nursing care requiring insulin therapy.

GlucoTab has a CE certificate, will be used according to its intended purpose and no additional burdensome or invasive interventions are planned

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained after being advised of the nature of the study
* Male or female aged ≥ 18 years
* Type 2 diabetes (treated with insulin therapy)
* Receiving domiciliary nursing care

Exclusion Criteria:

* type 1 diabetes mellitus
* intravenous insulin therapy
* hyperglycaemic episodes (ketoacidosis, hyperosmolar state) if they require intravenous insulin therapy
* continuous subcutaneous insulin infusion
* gestational diabetes or pregnancy
* known or suspected allergy to insulin
* total parenteral nutrition
* any mental condition rendering the patient incapable of giving his/her consent
* any disease or condition which according to the investigator would interfere with the trial or the safety of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-critically ill patients with type 2 diabetes receiving domiciliary nursing care who require s.c. insulin therapy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-11-30 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Efficacy - mean percentage of Fasting Blood Glucose | ≥ 24 hours after start of the therapy by using the GlucoTab system
  Efficacy is assessed by evaluating the mean percentage of Fasting Blood Glucose (FBG) in the FBG target range 80 - 180 mg/dl

SECONDARY OUTCOMES:
Safety - number of hypoglycaemic events | at the end of the study, on average three months
  Safety is assessed by evaluating the number of hypoglycaemic events
Efficacy - mean pre-breakfast blood glucose values | at the end of the study, on average three months
  Efficacy is further assessed by the measurement of mean pre-breakfast blood glucose values
Usability | at the end of the study, on average three months
  Percentage of insulin dose injections performed according to the GlucoTab system

CONTACTS AND LOCATIONS:
Locations (1):
- Austrian Red Cross, Graz, Austria